CLINICAL TRIAL: NCT05032209
Title: Follow-up of Children With Severe Asthma at Adult Age
Acronym: S2AEA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP210852; IDRCB: 2021-A00825-36 (Other: ANSM)
Record Dates: First submitted 2021-08-27; First posted 2021-09-02 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Severe Asthma
Keywords: childhood; adulthood
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: follow-up of children with severe asthma in adulthood — follow-up of children with severe asthma in adulthood

SUMMARY:
Most of clinical cohorts focused on the course of asthma over time and on the different phenotypes of asthma have investigated children and adults separately. The passage from childhood to adulthood is scarcely explored.

In this context, we decided to explore the course of asthma severity from teenage to adulthood in children with severe asthma. The secondary objectives are to assess the quality of life and socioeconomic status in adulthood.

This study will be both retrospective (data collected during childhood) and prospective (data collected during adulthood), multicentric and observational

DETAILED DESCRIPTION:
Asthma is one of the most frequent pediatric chronic disease; between 30% and 50% of preschoolers have one to more episodes of wheezing, but less than half of them will have asthma persisting during childhood .Over the past decades, several longitudinal studies have described the different trajectories of asthma depending on the initial phenotype. The results of the MAS study (Melbourne Asthma Study), including 330 patients followed from the age of 7 to the age of 35 and then 50 years, showed that the most symptomatic asthma at school age was most at risk of persisting into adulthood. Risk factors for persisting symptomatic asthma were female gender, history of atopic dermatitis, changes in respiratory function in childhood, parental history of asthma, early onset of asthma, and frequency exacerbations in childhood. Thus, severe childhood asthma is more likely to persist in adulthood while mild asthma is more likely to go into remission. Long-term remission is still possible; in the MAS cohort, 15% of patients with severe childhood asthma were in complete remission by the age of 50 years.Severe asthma is poorly represented in studies from the general population or neonatal cohorts, as it remains rare in children. However, there are several clinical studies supporting at least a partial improvement in symptoms in adulthood. Thus, in a Dutch cohort of asthmatic children followed in a tertiary center and re-assessed in their 2nd and 3rd decades, asthma symptoms returned to at least partial remission in 52% of patients. However, only a minority of them (42%) had complete remission of their symptoms and normal respiratory function.Most of the clinical cohort studies examining the prognosis of asthma during time explored separately children and adults. Some biomarkers are lacking in children and the passage from childhood to adulthood is not explored. The usual phenotypic description takes into account the presence or absence of atopy, the frequency of symptoms, the factors triggering exacerbations, the severity of the disease, some biomarkers of inflammation and the level of control under treatment. The difficulty of accessing biomarkers from the deep lung in children and the binary analysis of some variables such as atopy make the description and the analysis of risk factors for persistence of asthma in adulthood difficult.

In addition, the prognosis of asthma is not only influenced by biological and environmental factors, but also by social factors throughout life. Thus, a low socioeconomic level is a recognized risk factor for severe acute asthma and poor asthma control.Finally, beyond the medium and long term prognosis, severe asthma is associated with an impaired quality of life, in children as well as in adults.In this context, the main objective of this study is to determine the course of asthma from childhood to young adulthood in a population of children with severe persistent asthma. The secondary objectives are to determine the phenotypic evolution of asthma (in particular atopic co-morbidities); to Compare the severity of asthma in adulthood according to the initial phenotypes of asthma in childhood, integrating clinical, functional, radiological, and biological parameters (including biomarkers from the deep lung);to describe the quality of life of these patients in adulthood and their socio-economic status.The primary endpoint is the classification of the severity and control of asthma in adulthood according to the GINA criteria.The secondary endpoints will be :

- When assessing severe asthma in childhood: Demographic data: age, sex, term of birth, socio-economic level of parents according to INSEE (high, intermediate or low), geographic origin of parents, body mass index.

Environmental data: exposure to irritants and potential allergens. Anamnestic data: history of familial asthma, time to disease progression, history of pneumonia, bronchopulmonary dysplasia.

Associated co-morbidities: existence of allergic rhinitis assessed by the SFAR diagnostic score and the ARIA severity score, atopic dermatitis, food allergy, clinical gastroesophageal reflux disease or proven by pHmetry.

Results of additional assessments: bronchial endoscopy, functional respiratory data, blood eosinophilia, existence of allergen sensitization

During Adulthood :

Demographic data: age at time of collection, BMI. Social data: level of education, socio-professional category according to INSEE, disability, health insurance, number of days of school or professional absenteeism for asthma out of the 12 last months.

Environmental data: exposure to irritants and potential allergens. Associated co-morbidities: allergic rhinitis assessed by the SFAR diagnostic score and the ARIA severity score, atopic dermatitis, food allergy, gastroesophageal reflux disease Evaluation of the quality of life by the mini-AQLQ score. Results of additional examinations carried out in the year of the assessment: Respiratory functional data.

During Adulthood :

Demographic data: age at time of collection, BMI. Social data: level of education, socio-professional category according to INSEE, disability, health insurance, number of days of school or professional absenteeism for asthma out of the 12 last months.

Environmental data: exposure to irritants and potential allergens. Associated co-morbidities: allergic rhinitis assessed by the SFAR diagnostic score and the ARIA severity score, atopic dermatitis, food allergy, gastroesophageal reflux disease Evaluation of the quality of life by the mini-AQLQ score.

Results of additional examinations carried out in the year of the assessment: Respiratory functional data.Design of the study : Multicentric, observational, both retrospective and prospective study. Inclusion and non-inclusion criteria :

Inclusion criteria

* to be aged at least 18 years old in 2021
* Have had an evaluation for severe asthma during childhood at Trousseau Hospital or Robert Debré Hospital
* Affiliation to an health insurance coverage. Non-inclusion criteria
* Patient without severe asthma at the time of the assessment in childhood
* Patient with an associated respiratory disease other than asthma (bronchopulmonary dysplasia, cystic fibrosis, primary ciliary dyskinesia) whose diagnosis has been invalidated or confirmed during the initial assessment
* Patient opposition

ELIGIBILITY:
Inclusion Criteria:

* to be aged at least 18 years old in 2021
* Have had an evaluation for severe asthma during childhood at Trousseau Hospital or Robert Debré Hospital
* Affiliation to an health insurance coverage. Non-inclusion criteria

Exclusion Criteria:

* Patient without severe asthma at the time of the assessment in childhood
* Patient with an associated respiratory disease other than asthma (bronchopulmonary dysplasia, cystic fibrosis, primary ciliary dyskinesia) whose diagnosis has been invalidated or confirmed during the initial assessment
* Patient opposition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinical cohort of adults patients with severe asthma in childhood
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-07-12 (Actual); Primary Completion 2022-07-12 (Estimated); Study Completion 2022-07-12 (Estimated)

PRIMARY OUTCOMES:
severity and control of asthma in adulthood according to the GINA criteria | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Flore AMAT, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Robert Debre Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided